CLINICAL TRIAL: NCT05581147
Title: Thyroid Function and Structure in Klinefelter Syndrome (THINKS)
Brief Title: Thyroid Function and Structure in Klinefelter Syndrome
Acronym: THINKS
Status: Recruiting | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Andrea M. Isidori, Full professor, University of Roma La Sapienza
Other Study IDs: THINKS
Record Dates: First submitted 2022-10-04; First posted 2022-10-14 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-02

CONDITIONS: Klinefelter Syndrome; Thyroiditis, Autoimmune; Hypothyroidism
Keywords: Klinefelter syndrome; Hypothyroidism; Thyroiditis; Puberty; Prepuberty; Testosterone
MeSH Terms: conditions — Klinefelter Syndrome; Thyroiditis, Autoimmune; Hypothyroidism; Thyroiditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Klinefelter syndrome: Males affected by 47,XXY non-mosaic Klinefelter syndrome. Subgroups according to pubertal stage: pre-pubertal, pubertal and adults. Subgroups according to gonadal status: eugonadal, hypogonadal and receiving testosterone replacement therapy (TRT).
- Healthy controls: Euthyroid, age- and pubertal stage-matched males Subgroups according to pubertal stage: pre-pubertal, pubertal and adults.
- Chronic lymphocytic thyroiditis: Adult males affected by chronic lymphocytic thyroiditis

SUMMARY:
This is a longitudinal retrospective study for the evaluation of thyroid function and structure in patients with Klinefelter syndrome compared to healthy controls and patients affected by chronic lymphocytic thyroiditis.

DETAILED DESCRIPTION:
This is a longitudinal retrospective study for the evaluation of thyroid function and structure in patients with Klinefelter syndrome compared to healthy controls and patients affected by chronic lymphocytic thyroiditis (CLT).

The investigators will retrospectively enroll patients with Klinefelter syndrome followed at the host institution and will retrieve data with regards to peripheral hormone levels (thyroid function) and ultrasonographic appearance (thyroid structure) according to pubertal status and gonadal status. Data will be compared with male age- and pubertal stage-matched euthyroid controls, as well as with male patients affected by CLT.

The primary outcome will be the thyroid function compared to healthy controls, by the assessment of peripheral blood TSH, free T3 (fT3) and free T4 (fT4) levels according to pubertal status (pre-pubertal, pubertal and adult subjects) as well as according to gonadal status (eugonadal subjects, hypogonadal subjects and subjects receiving testosterone replacement therapy [TRT]).

Secondary Outcome Measures will be:

Thyroid function indexes (fT3/fT4 ratio, fT4/TSH ratio, TSH*fT4 product)

Quantitative ultrasonographic thyroid structure parameters, comprising: thyroid volume and echogenicity index, as well as the echotexture parameters of homogeneity and entropy evaluated by Gray Levels Co-occurrence Matrices (GLCM).

In vitro assay of testosterone and estradiol effects on deiodinase type 2 (DIO2) activity in a rat pituitary cell line.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of classic, non-mosaic 47,XXY Klinefelter syndrome based on a peripheral blood 97 karyotype analysis;
* Availability of thyroid function test results (TSH, fT3, and fT4) and/or thyroid US imaging;
* Availability of concurrent clinical data.

Exclusion Criteria:

* Presence of other known genetic conditions or chromosomal abnormalities;
* Use of levothyroxine or other drugs that are either active on the hypothalamic-pituitary-thyroid (HPT) axis or that may interfere with thyroid function tests;
* History of previous surgery or radiotherapy on the thyroid or pituitary glands;
* Current or previous T therapy (for the pre-pubertal and pubertal groups).

Ages: 1 Year to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will enroll three cohorts of patients:
  * Patients with a confirmed diagnosis of classic, non-mosaic 47,XXY Klinefelter syndrome;
  * Males with a diagnosis of chronic lymphocytic thyroiditis (CLT); adult male patients affected by CLT, defined by positivity to anti-thyroglobulin antibodies (Ab-Tg) and/or anti-thyroperoxidase antibodies (Ab-TPO);
  * Euthyroid, healthy controls with no clinical signs or symptoms of thyroidal or testicular disease and meeting the same inclusion and exclusion criteria described above (except for KS diagnosis and availability of thyroid US in pre-pubertal and pubertal children).
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2007-05-11 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Peripheral blood TSH concentration | Through study completion, an average of 6 years
  Thyroid function will be assessed by peripheral blood TSH levels, taking into account pubertal status (pre-pubertal, pubertal and adult subjects) as well as to gonadal status (eugonadal subjects, hypogonadal subjects and subjects receiving TRT).
Peripheral blood fT3 concentration | Through study completion, an average of 6 years
  Thyroid function will be assessed by peripheral blood free T3 (fT3) levels, taking into account pubertal status (pre-pubertal, pubertal and adult subjects) as well as to gonadal status (eugonadal subjects, hypogonadal subjects and subjects receiving TRT).
Peripheral blood fT4 concentration | Through study completion, an average of 6 years
  Thyroid function will be assessed by peripheral blood free T4 (fT4) levels, taking into account pubertal status (pre-pubertal, pubertal and adult subjects) as well as to gonadal status (eugonadal subjects, hypogonadal subjects and subjects receiving TRT).

SECONDARY OUTCOMES:
Peripheral deiodinase 2 (DIO2) activity | Through study completion, an average of 6 years
  The investigators will derive the the fT3/fT4 ratio as a surrogate marker of peripheral deiodinase 2 (DIO2) activity.
Pituitary sensitivity sensitivity to thyroid hormones | Through study completion, an average of 6 years
  The investigators will derive the fT4/TSH ratio as surrogate marker of pituitary sensitivity.
Thyroid hormone resistance index | Through study completion, an average of 6 years
  The investigators will derive the TSH*fT4 product as a surrogate marker of thyroid hormone resistance.
Thyroid volume | Through study completion, an average of 6 years
  The investigators will assess ultrasonography-derived thyroid volume (in mL) by the sum of the left and right lobe volumes, derived by the ellissoid formula (d1 x d2 x d3 x 0,5233).
Quantitative thyroid echogenicity | Through study completion, an average of 6 years
  The investigators will assess the ultraonographic thyroid echogenicity index, derived by the histogram mean of thyroid parenchyma in a standardized scan, normalized by the histogram mean of the pre-thyroid muscles.
Thyroid echotexture (homogeneity) | Through study completion, an average of 6 years
  The investigators will assess the ultrasonographic thyroid parenchymal echotexture via the analysis of Grey Levels Co-occurrence Matrices (GLCM) second-order parameter homogeneity (or IDM).
Thyroid echotexture (entropy) | Through study completion, an average of 6 years
  The investigators will assess the ultrasonographic thyroid parenchymal echotexture via the analysis of Grey Levels Co-occurrence Matrices (GLCM) second-order parameter entropy.
In vitro assay of deiodinase type 2 (DIO2) activity | At study end (May 2022).
  The investigators will assess in vitro modulation of DIO2 activity by sex hormones testosterone and 17-beta estradiol in a rat pituitary cell line (GH4C1) by using a thyroid hormone-responsive artificial promoter (TRE3Tk-Luc).

CONTACTS AND LOCATIONS:
Overall Officials: Andrea M Isidori, MD, PhD, Principal Investigator — andrea.isidori@uniroma1.it
Locations (1):
- 'Sapienza' University of Rome, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided